CLINICAL TRIAL: NCT06908733
Title: Prognosis and Patient-Reported Outcomes of Combined Local Treatments (Surgery and Radiotherapy or Radiotherapy Alone) With Tislelizumab and Chemotherapy in Initial Stage III-N3 Non-Small Cell Lung Cancer: A Prospective, Open-Label, Single-Arm, Phase II Trial
Brief Title: Integrating Surgery and Radiotherapy Following Tislelizumab-based Conversion Therapy in N3-Stage III NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HURRICANE (LCH-LT04)
Record Dates: First submitted 2025-03-12; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer (Stage III)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab + Chemotherapy +Local Treatments (Surgery and Radiotherapy or Radiotherapy Alone) (Experimental): Following induction therapy with 3-4 cycles of Tislelizumab combined with platinum-based chemotherapy, patients without disease progression will be evaluated by a multidisciplinary team (MDT) and assigned to treatment strategies based on eligibility and patient preference. Patients deemed eligible to surgery will receive standard lung cancer resection (excluding total pneumonectomy), including removal of the primary tumor, ipsilateral hilar, and ipsilateral mediastinal lymph nodes, followed by hypofractionated chemoradiotherapy targeting N3 metastatic lymph nodes. Patients ineligible for or unwilling to undergo surgery will receive definitive conventional CRT. After completion of local treatment, all patients will continue Tislelizumab maintenance therapy until radiographic disease progression, unacceptable toxicity, or completion of one year of treatment.
  Interventions: Drug: 3-4 cycles of Tislelizumab combined with platinum-based chemotherapy, evaluated by MDT and assigned to treatment strategies based on eligibility and patient preference.

INTERVENTIONS:
Drug: 3-4 cycles of Tislelizumab combined with platinum-based chemotherapy, evaluated by MDT and assigned to treatment strategies based on eligibility and patient preference. — Patients deemed eligible to surgery will receive standard lung cancer resection (excluding total pneumonectomy)

SUMMARY:
This is a prospective, open, multicenter, Phase II single-arm clinical study. In subjects with an initial stage of stage III-N3 non-small cell lung cancer (NSCLC) that was negative for sensitive gene mutations and had not received any systemic or local therapy (T1-4N3M0, excluding primary tumor or metastatic lymph node invasion of the aorta/trachea/esophagus/heart, etc.); After 3-4 cycles of Tislelizumab combined with platinum-containing dual agents, the patients without disease progression were evaluated by MDT and selected according to the patient's wishes, including those who could receive conventional/standard radical lung cancer surgery (excluding total lung resection). Conventional/standard resection of primary, ipsilateral hilum and ipsilateral mediastinum combined with hypofractionted chemoradiotherapy of N3 metastatic lymph nodes was performed. For patients who are inoperable or unwilling to undergo surgery or intolerant to surgery, conventional concurrent chemoradiotherapy is given. Maintenance therapy with Tislelizumab was continued after local treatment until disease progression, drug intolerance as assessed by imaging, or after 1 year; Participants were followed up according to the procedure to evaluate efficacy and patient-reported outcomes.

The study included a screening period (no more than 28 days after subjects signed informed consent to the first dose), a treatment period (including Tislelizumab combined with chemotherapy-restaging and MDT-local treatment-maintenance therapy), and a follow-up period.

Thirty patients：30 patients Primary endpoint: 1-year EFS rate Secondary endpoints: EFS, OS, surgical rate, TTDM, TTLR, AEs, PROs Exploratory end points: Imaging efficacy, pathological efficacy and other relevant clinical outcomes; Predictive biomarkers based on tissue and blood samples.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single arm phase 2 clinical trial enrolling 30 newly diagnosed stage III NSCLC patients with N3 lymph-node metastasis (T1-4N3M0, AJCC 9th edition). Mainly eligible patients must be negative for sensitive gene muta-tions, treatment-naive for systemic or local therapy, aged ≥18 years, and have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, with at least one measurable lesion according to RECIST 1.1 criteria at baseline. Key exclu-sion criteria include invasion of critical structures such as the aorta, trachea, esopha-gus, or heart by the primary tumor or metastatic lymph nodes, as well as the presence of Pancoast tumors. Following induction therapy with 3-4 cycles of Tislelizumab combined with platinum-based chemotherapy, patients without disease progression will be evaluated by a multidisciplinary team (MDT) and assigned to treatment strategies based on eligibility and patient preference. Patients deemed eligible to surgery will receive standard lung cancer resection (excluding total pneumonectomy), including removal of the primary tumor, ipsilateral hilar, and ipsilateral mediastinal lymph nodes, followed by hypofractionated chemoradiotherapy targeting N3 meta-static lymph nodes. Patients ineligible for or unwilling to undergo surgery will re-ceive definitive conventional CRT. After completion of local treatment, all patients will continue Tislelizumab maintenance therapy until radiographic disease progres-sion, unacceptable toxicity, or completion of one year of treatment. The primary endpoint is the 1-year event-free survival rate (1y-EFS rate). Secondary endpoints include EFS, overall survival (OS), surgical conversion rate, time to distant metasta-sis (TTDM), time to local recurrence (TTLR), adverse events (AEs), and the impact of the integrated treatment approach on patient-reported outcomes (PROs). Explora-tory analyses will be conducted to identify predictive and prognostic biomarkers us-ing tumor tissue and blood samples collected at multiple time points during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older (inclusive);
2. Willingness to participate and provide written informed consent;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1, with no deterioration in the two weeks prior to treatment, and an expected survival of at least 12 weeks;
4. Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), T1-4N3M0 (AJCC 9th edition); suspicious lymph nodes on whole-body 18F-fluorodeoxyglucose positron emission tomography (PET) or contrast-enhanced computed tomography (CT) or PET-CT should undergo invasive lymph node staging which can be confirmed through endobronchial ultrasound, mediastinoscopy, thoracoscopy, or needle biopsy; however, mandatory confirmation is not required for highly suspicious mediastinal lymph nodes in zones 5 and 6;
5. For patients with non-squamous cell carcinoma, EGFR, ALK, etc., testing results based on tumor tissue or blood samples must be provided; for squamous NSCLC patients, if the sensitive gene mutation status is unknown, it is not required to perform such tests during screening;
6. No prior systemic therapy or local treatment after diagnosis of NSCLC;
7. At least one measurable lesion according to RECIST 1.1 criteria at baseline. The longest diameter should be ≥10 mm (if a lymph node, the shortest diameter should be ≥15 mm). The chosen method of measurement should be suitable for accurate repeated measurements, such as CT or MRI. If only one measurable lesion exists, it may be accepted as the target lesion, evaluated at least 14 days after diagnostic biopsy. Baseline imaging assessment should be performed within 28 days before the first dose of study medication;
8. Women of childbearing potential must use effective contraception from screening until six months after discontinuation of study treatment and should not breastfeed. Prior to starting treatment, a negative pregnancy test is required, or one of the following criteria proving no risk of pregnancy: ① Postmenopausal defined as age greater than 50 years and amenorrhea for at least 12 months following cessation of all exogenous hormonal replacement therapy; ② Women under 50 years old who have been amenorrheic for 12 months or more after stopping all exogenous hormonal therapy and whose levels of luteinizing hormone (LH) and follicle-stimulating hormone (FSH) fall within laboratory postmenopausal reference ranges are also considered postmenopausal; ③ History of irreversible sterilization surgery including hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not bilateral tubal ligation;
9. Non-sterilized males must use barrier contraception (i.e., condoms) from screening until six months after discontinuation of study treatment; sterilized males are defined as: a. Males with azoospermia confirmed by semen sample examination prior to the study, serving as definitive evidence of male sterilization; b. In this study, males known to have "low sperm count" (meeting the definition of "subfertility") are still considered fertile and not infertile.

Exclusion Criteria:

1. Diagnosed with Pancoast tumor;
2. Pathologically confirmed large cell neuroendocrine carcinoma (LCNEC);
3. Primary tumor or metastatic lymph nodes infiltrating major vessels/aorta, trachea, esophagus, heart, etc.;
4. Any of the following prior treatments: ① Previous lung surgery; ② Prior systemic chemotherapy, immunotherapy, targeted therapy, or any other anti-tumor treatment for lung cancer; ③ Known presence of epidermal growth factor receptor (EGFR) mutations, ALK rearrangements, ROS1 rearrangements, BRAF V600 mutations, RET rearrangements, MET exon 14 skipping mutations, NTRK1/2/3 rearrangements, or other sensitive mutations; ④ Prior radiotherapy to the lungs; ⑤ Major surgery within 14 days prior to first dose or within 28 days if not fully recovered from toxicity and/or complications; ⑥ Use of traditional Chinese medicine with anti-tumor effects is allowed if discontinued at least 2 weeks before study drug administration and used for no more than 7 days;
5. Diagnosis of other malignancies within the last 5 years, except for completely resected basal cell or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix, or breast carcinoma in situ;
6. Active autoimmune disease or history of autoimmune disease that may recur [excluding patients with well-controlled type 1 diabetes, hypothyroidism (if controlled by hormone replacement therapy alone), celiac disease, non-systemic dermatological conditions (e.g., vitiligo, psoriasis, alopecia), or any other disease not expected to recur without external triggers];
7. Conditions requiring systemic corticosteroid therapy (> 10 mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days prior to first dose [patients currently or previously using any of the following steroid regimens are eligible: adrenal replacement steroids (prednisone ≤ 10 mg/day or equivalent), minimal systemic absorption of local, ocular, intra-articular, intranasal, and inhaled corticosteroids, short-term (≤ 7 days) use of corticosteroids for prophylaxis or treatment of non-autoimmune conditions];
8. Uncontrolled diabetes or laboratory abnormalities (> Grade 1) in potassium, sodium, or corrected calcium despite standard medical management within 14 days prior to first dose;
9. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring frequent drainage (recurrence within 2 weeks after intervention);
10. History of interstitial lung disease or active interstitial lung disease, pneumonitis (non-infectious), or uncontrolled pulmonary conditions (e.g., pulmonary fibrosis, acute interstitial lung disease);
11. Fever ≥ 38°C within 7 days prior to first dose, significant active infection, active tuberculosis, or active fungal, bacterial, or viral infections requiring systemic treatment [chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection patients receiving antiviral therapy are allowed];
12. Untreated chronic hepatitis B or chronic HBV carriers with HBV DNA > 500 IU/mL (or > 2500 copies/mL) [inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B patients (HBV DNA < 500 IU/mL or < 2500 copies/mL) are eligible. Patients with detectable HBsAg or HBV DNA should be managed according to guidelines];
13. Active HCV infection [patients with negative HCV antibody tests or positive HCV antibody but negative HCV RNA tests are eligible. Only patients with positive HCV antibody tests will undergo HCV RNA testing];
14. Known history of HIV infection;
15. Prior allogeneic stem cell transplantation or organ transplantation;
16. Any cardiovascular risk factors: ① Cardiac chest pain within 28 days prior to first dose; ② Pulmonary embolism within 28 days prior to first dose; ③ Acute myocardial infarction within 6 months prior to first dose; ④ NYHA Class III or IV heart failure within 6 months prior to first dose; ⑤ ≥ Grade 2 ventricular arrhythmia within 6 months prior to first dose; ⑥ Cerebrovascular accident within 6 months prior to first dose; ⑦ Uncontrolled hypertension (≥ CTCAE Grade 3) despite medication within 28 days prior to first dose; ⑧ Syncope or seizure within 28 days prior to first dose; ⑨ Left ventricular ejection fraction (LVEF) ≤ 40% [patients with coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF between 40% and 50% must receive optimized stable treatment as per their physician's advice, consulting a cardiologist if necessary];
17. History of severe hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins;
18. Allergy to pemetrexed, its excipients, cisplatin/carboplatin, albumin-bound paclitaxel, or other platinum compounds; contraindications to cisplatin such as hearing impairment;
19. Severe or uncontrolled systemic diseases, unstable or uncompensated respiratory, hepatic, or renal diseases;
20. Insufficient bone marrow reserve or organ function, meeting any of the following laboratory limits (without corrective treatment within one week prior to blood draw): ① Absolute neutrophil count < 1.5 × 10^9/L; ② Platelet count < 90 × 10^9/L; ③ Hemoglobin < 90 g/L (< 9 g/dL); ④ Alanine aminotransferase > 2.5 × ULN; ⑤ Aspartate aminotransferase > 2.5 × ULN; ⑥ Total bilirubin > 1.5 × ULN (Gilbert syndrome allowed); ⑦ Creatinine > 1.5 × ULN (confirmation of creatinine clearance required); ⑧ Serum albumin (ALB) < 25 g/L; ⑨ INR or aPTT > 1.5 × ULN for patients not on anticoagulant therapy;
21. Any immunotherapy (e.g., interleukins, interferons, thymosin, etc.) or experimental treatment within 14 days or 5 half-lives (whichever is longer) prior to first dose;
22. Live vaccines or live-attenuated vaccines within 28 days prior to first dose [seasonal influenza vaccines are generally inactivated and allowed; intranasal vaccines are live and not allowed];
23. Underlying diseases (including laboratory abnormalities), alcohol or drug abuse, or dependence that could interfere with study treatment administration, toxicity assessment, adverse event interpretation, or reduce compliance with the study protocol;
24. Concurrent participation in another therapeutic clinical trial [concurrent participation in observational or non-interventional studies is allowed];
25. Pregnant, lactating, or planning to become pregnant during the study period;
26. Participants judged by the investigator to have poor compliance with study procedures and requirements due to a history of neurological or psychiatric disorders (including epilepsy or dementia), current mental health conditions, etc.;
27. Participants deemed by the investigator to have any condition that endangers safety or interferes with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
1-year EFS rate | treatment period：Induction therapy (Day 1 of medication); Surgery+Radiotherapy/Radiotherapy; maintenance therapy (one year). follow-up period：One year after the completion of maintenance therapy (one year).
  The 1-year Event-Free Survival (EFS) rate is defined as the proportion of patients who have not experienced an EFS event at one year after the first administration of the study drug. EFS is defined as the time from the first dose of the study treatment until the first objective documentation of disease progression that renders the patient unresectable or ineligible for curative radiotherapy, local recurrence, distant metastasis, or death from any cause, whichever occurs first. EFS is assessed by the investigator based on RECIST v1.1 criteria using the curative intent treatment analysis set.

SECONDARY OUTCOMES:
Secondary endpoints: EFS, OS, surgical rate, TTDM, TTLR, AEs, PROs | treatment period：Induction therapy (Day 1 of medication); Surgery+Radiotherapy/Radiotherapy; maintenance therapy (one year). follow-up period：One year after the completion of maintenance therapy (one year).
  OS: The duration from study enrollment to death from any cause. Surgical rate: Percentage of operable patients receiving surgical resection. TTDM: The percentage of patients from enrollment to the first detection of tumor metastasis in distant organs or tissues compared to the number of patients in the corresponding treatment group.
  TTLR: The percentage of patients with tumor recurrence at the primary lesion or adjacent area after treatment compared to the number of patients in the corresponding treatment group.
  AEs: Classify and grade adverse events according to the latest version of the Common Terminology Criteria for Adverse Events (CTCAE), and assess the incidence, severity, and causal relationship of treatment-related adverse events.
  PROs: Collect data directly from patients regarding their health status or treatment impact using specific tools (such as FACT-G), without interpretation by healthcare professionals, to provide a patient perspective on treatment effects.